CLINICAL TRIAL: NCT00688974
Title: Longitudinal Cohort Study Comparing 2 Surgical Techniques (Roux-en-Y Gastric Bypass and Adjustable Gastric Banding) in Patients With Class 3 Obesity and Type 2 Diabetes
Brief Title: Longitudinal Cohort Study Comparing 2 Surgical Techniques in Patients With Class 3 Obesity and Type 2 Diabetes
Acronym: OBEDIAB
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: DGS 2004/0123; 2004/0412 (Other: sponsor)
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: type 2 diabetes; obesity; gastric bypass; adjustable gastric banding; BMI > 35.; obesity for more than 5 years
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma during meal test (0, 30, 60, 90, 120, 180 min)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Roux-en-Y gastric bypass: Patients with class 3 obesity and type 2 diabetes submitted to Roux-en-Y gastric bypass
  Interventions: Procedure: Roux-en-Y gastric bypass
- Adjustable gastric banding: Patients with class 3 obesity and type 2 diabetes submitted to adjustable gastric banding
  Interventions: Procedure: Adjustable gastric band
- Healthy controls: Non-obese, non-diabetic adults

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass — Laparoscopic Roux-en-Y gastric bypass
  Other Names: Gastric bypass
  Groups: Roux-en-Y gastric bypass
Procedure: Adjustable gastric band — Laparoscopic adjustable gastric band
  Other Names: Gastric Banding
  Groups: Adjustable gastric banding

SUMMARY:
Wight loss surgery provides good glycemic control in type 2 diabetes. The technique of "Roux-en-Y gastric bypass" is more effective than the "Adjustable Gastric Band" on weight loss.

This longitudinal cohort study will compare the effectiveness of the Roux-en-Y gastric bypass and Adjustable Gastric Banding on glycemic control in type 2 diabetes and explore the responsible mechanisms.

The evaluation will be made preoperatively and 1 year later as assessed by the decline in HbA1c. An evaluation will also be carried out after a weight loss of 10% to indicate whether the observed difference is independent of weight loss.

DETAILED DESCRIPTION:
Type 2 diabetes is a condition often associated with obesity and often difficult to control. In patients with severe obesity, surgical treatment allows a sustainable weight loss and higher than that obtained with other treatments available. In most cases, surgery also reduces significantly the comorbidities of obesity and diabetes in particular. Among the various technical options, adjustable gastric band (AGB) is the simplest and by far the most used in France.

Roux-en-Y gastric bypass (RYGB) is a more complicated intervention combining gastrointestinal malabsorption- duodeno-jejunal and gastric reduction and allows a higher weight loss. Several studies also suggest that the technique has a remarkable efficiency on glycemic control, justifying the extension of its readings/indications. No study controlled, however, has compared these two techniques.

The objective of this study is to compare the efficiency of RYGB vs AGB on glycemic control in type 2 diabetes. Although some studies have compared AGB and RYGB, none have compared their effectiveness on post prandial glucose control in patients with diabetes. It is generally recognized that the effectiveness of RYGB on diabetes is independent of the weight loss, but this has never been demonstrated.

By demonstrating the superiority of RYGB vs AGB, and identifying the responsible mechanisms, the study will expand the indications of RYGB in the treatment of type 2 diabetes. Weight loss surgery offers a unique model for the clinical study of the pathophysiology of type 2 diabetes.

Main objective:

* To compare the effectiveness of RYGB vs AGB on glucose control in obese patients with type 2 diabetes.

Secondary Objectives:

* demonstrate that the better outcome achieved with RYGB is independent of weight loss.
* Identify the mechanisms underlying the better outcome of RYGB

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years AND
* BMI > 35
* Type 2 diabetes
* Obesity for more than 5 years OR
* normoglycemia
* BMI< 30

Exclusion Criteria:

* Secondary obesity due to an endocrinopathy
* Chronic pathology (neoplasia, cirrhosis, disease of system)
* Psychosis, alcoholic addiction or narcotics.
* Contre-indications to the anaesthesia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Candidate for bariatric surgery (Roux-en-Y gastric bypass OR adjustable gastric band) with class 3 obesity (body mass index ≥ 35 kg/m2) and type 2 diabetes (ADA definition)
  OR healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2004-05; Primary Completion 2006-11 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Glucose control | 12 months
  HbA1c and fasting blood glucose

SECONDARY OUTCOMES:
Glycaemia, Insulinemia, Incretins during a standardized meal test at 10% of weight loss | 3 months
  Concentration curves of glycaemia, insulinemia, incretins, and D-xylose during a standardized mixed meal test
Weight loss | 60 months
  Body mass index
Glycaemia, Insulinemia, Incretins, and D-xylose during a normalized(standardized) meal | 12 months
  Concentration curves of glycaemia, insulinemia, incretins, and D-xylose during a standardized mixed meal test
Glycaemia, insulinemia, incretins, and D-xylose during a normalized(standardized) meal | 60 months
  Concentration curves of glycaemia, insulinemia, incretins, and D-xylose during a standardized mixed meal test
Diabetes remission | 60 months
  HbA1c < 6.5% AND fasting blood glucose < 7.0 mmol/L in absence of antidiabetic drug

CONTACTS AND LOCATIONS:
Overall Officials: Francois PATTOU, Principal Investigator — Lille University Hospital
Locations (1):
- Lille University Hospital, Lille, Nord, France